CLINICAL TRIAL: NCT06232824
Title: Multicomponent Supervised Tele-rehabilitation Versus Home-based Self-rehabilitation After Anterior Cruciate Ligament Reconstruction
Brief Title: Tele-rehabilitation After Anterior Cruciate Ligament Reconstruction
Acronym: tele-rehab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kexin Wang, MM (Other)
Responsible Party: Sponsor-Investigator, Kexin Wang, MM, Clinical Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WestChinaH20240116
Record Dates: First submitted 2024-01-16; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Tele-rehabilitation; Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Intervention Participants in the intervention group coud only view the rehabilitation content that needs to be carried out at the current phase every day and confirm whether to execute it on the application. Participants could communicate with therapists on the mobile phone application by sending text, voice, images, and videos throughout the entire experiment.
  Control Participants in the control group could only receive a graphic and textual minimal postoperative rehabilitation plan on the mobile phone application. However, the participants was not informed the frequency and intensity of the rehabilitation items. They could not communicate with therapists online. Participants in the control group was expected to exercise unsupervised postoperatively.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded participants and therapists were not implemented in our study. Before the intervention, an independent researcher communicated with the patient to inform the method of using the mobile application. Apart from the mobile application, no paper rehabilitation program materials will be distributed to participants. Admission, ACLR surgery, follow-up, and assessment of all participants were conducted separately and will not be arranged in the same ward room to avoid discussion and communication between participants. The ACLR surgery was performed by a senior surgeon who was blinded to the group allocation. In addition, we selected two assessors who were blinded to the group allocation to measure the baseline data and follow-up outcomes after the intervention. The collection and analysis of data were carried out by two independent researchers who were also blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group coud only view the rehabilitation content that needs to be carried out at the current phase every day and confirm whether to execute it on the application. Participants could communicate with therapists on the mobile phone application by sending text, voice, images, and videos throughout the entire experiment.
  Participants in the intervention group received detailed education and rehabilitation program on the mobile phone application including text, photos, and videos. On the first day of enrollment, the doctor inform the participants of the importance of rehabilitation and how to use the mobile phone application. The postoperative rehabilitation protocol includes four phases: Phase 1 (0-2 weeks), Phase 2 (3-4 weeks), Phase 3 (5-8 weeks), Phase 4 (9-12 weeks), and Phase 5 (after 13 weeks).
  Interventions: Behavioral: Tele-rehabilitation
- Control (No Intervention): Participants in the control group could only receive a graphic and textual minimal postoperative rehabilitation plan on the mobile phone application. However, the participants was not informed the frequency and intensity of the rehabilitation items. They could not communicate with therapists online. Participants in the control group was expected to exercise unsupervised postoperatively.
  At the 2, 4, 8, 12, and 24 weeks after ACLR, all participants went to the outpatient clinic for follow-up by physiotherapist to provide face-to-face guidance for exercise methods. Physiotherapist would clarify the content of the rehabilitation plan if any doubt, but will not provide information extending the prearranged scope.

INTERVENTIONS:
Behavioral: Tele-rehabilitation — The whole program is constituted of preoperative education and postoperative rehabilitation (in hospital and out of hospital). All the participants received the same preoperative education through the mobile phone application and oral communication. Participants in the intervention group get the multicomponent supervised tele-rehabilitation, while participants in the control group get the home-based self-rehabilitation. All the postoperative rehabilitation programs are presented and executed through the mobile phone application.
  Arms: Intervention

SUMMARY:
The investigators aims to evaluate the effect of multicomponent supervised tele-rehabilitation, compared to home-based self-rehabilitation, on range of motion (ROM), pain, muscle strength, and function in patients following ACLR. The hypothesis is of superiority for the effects of multicomponent supervised tele-rehabilitation over home-based self-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 50 years at the time of recruit;
2. BMI between 16 and 28 kg/m²;
3. acute unilateral ACL rupture;
4. plan for an ACLR surgery (with autologous hamstrings tendon reconstruction) under arthroscopy;
5. ACL rupture to ACLR within 3 months;
6. Patients can independently use mobile software and WeChat mini programs, and can operate related software through the "Huajiantong" mini program under the guidance of staff;

Exclusion Criteria:

1. With synthetic tendon reconstruction;
2. Concomitant meniscus lesion which needs operation;
3. Concomitant other ligaments injury which needs operation;
4. Concomitant intra-articular knee fracture;
5. Concomitant fracture or injury which may affect postoperative exercise;
6. Previous history of knee infection, fracture, and surgery;
7. Participate in knee exercises and/or rehabilitation programs in the past three months;
8. Living outside the city, regular return to the hospital for follow-up cannot be guaranteed;
9. Serious cardiopulmonary disease and unable to participate in rehabilitation exercise;
10. Other reasons for exclusion (mental disorders, stroke, pregnancy, etc).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients who achieve a satisfactory active ROM (flexion and extension) | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  In the first 3 months after ACLR, the achievement of acceptable knee active extension and flexion was regarded as what matters most for a successful recovery. A good knee active ROM could guarantee an expectedly continue improvement.

SECONDARY OUTCOMES:
active and passive ROM | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The active and passive ROM of the affected side knee
Visual analogue scale (VAS) | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The postoperative pain was measured with VAS. The VAS scale ranges from 0 to 10 points, 0 points represent no pain, while 10 points represent the worst imaginable pain. A higher VAS score mean a worse outcome.
Muscle strength | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The isokinetic concentric strength test was used to assess muscle strength. Isokinetic concentric extenso was the best rated with sufficient intrarater reliability and construct validity for the measurement of knee muscle strength
The 2000 International Knee Documentation Committee (IKDC) | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The 2000 International Knee Documentation Committee (IKDC) Subjective Knee Form is a patient-oriented questionnaire that assesses symptoms and function in daily living activities. Scores are obtained by summing the individual items and then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
knee injury and osteoarthritis outcome score (KOOS) | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
the Tegner activity scale | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  the Tegner activity scale is a one-item questionnaire that is scored on an 11-item scale (0 to 10) based on the patient's reported level of activity/work. A level of 0 represents maximum disability while a level of 10 represents elite sports athletes.
the Lysholm knee scoring scale | at the 2, 4, 8, 12 and 24 weeks following the ACLR
  The Lysholm Knee Score is a questionnaire consisting of 8 items that the patient completes together with the therapist. The questionnaire is designed to assess the degree of knee instability at both impairment and limitation levels. .The Lysholm Knee Score calculates and grades an overall score from 0 to 100 based on 8 domains: squatting, locking, pain, stair climbing, support, instability, and edema.A higher score mean a better outcome. Scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang K, Peng L, You M, Deng Q, Li J. Multicomponent supervised tele-rehabilitation versus home-based self-rehabilitation management after anterior cruciate ligament reconstruction: a study protocol for a randomized controlled trial. J Orthop Surg Res. 2024 Jun 28;19(1):381. doi: 10.1186/s13018-024-04871-0. PMID 38943178